CLINICAL TRIAL: NCT06144203
Title: The Influence of Aerobic Exercise on Consolidation of Fear Extinction Learning in PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Principal Investigator, Kevin Crombie, Assistant Professor, University of Alabama, Tuscaloosa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: K01MH132545 (NIH)
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light-intensity aerobic exercise (Experimental)
  Interventions: Behavioral: Exercise
- Moderate-intensity aerobic exercise (Experimental)
  Interventions: Behavioral: Exercise
- High-intensity aerobic exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will complete either a 30-minute bout of light-, moderate-, or high-intensity aerobic exercise at one of the visits.

SUMMARY:
This study aims to test whether aerobic exercise performed after fear extinction learning improves cognitive, physiological, and neural indices of extinction recall in a sample of trauma-exposed men and women with and without posttraumatic stress disorder (PTSD). Participants will complete a clinical intake visit (Day 0), followed by a three-day fear conditioning (day 1), fear extinction + activity (day 2), and fear extinction recall (day 3) protocol.

ELIGIBILITY:
Inclusion Criteria for PTSD:

* male or female sex
* right-handed
* age 18-64
* a current diagnosis of PTSD where the index event involves interpersonal violence exposure (e.g., physical/sexual assault).

Inclusion criteria for the trauma-exposed (without PTSD) control participants includes:

* male or female sex
* right-handed
* age 18-64
* interpersonal violence exposure (e.g., physical/sexual assault).

Exclusion Criteria for all participants:

* current substance use disorder (other than alcohol, nicotine, or cannabis)
* acute suicidality
* history of bipolar/psychotic disorder
* changes to or addition of psychiatric medication in the past 4 weeks (6 weeks for fluoxetine)
* medications that effect neurovascular properties upon which BOLD fMRI capitalizes (e.g., water pills)
* history of neurological disorders or disease (e.g., traumatic brain injury, epilepsy, seizures)
* loss of consciousness > 10 minutes
* intellectual disabilities (IQ<70)
* developmental disorders
* MRI contraindication (e.g., internal ferromagnetic objects such as electronic devices, surgical implants, shrapnel; see phone screen)
* claustrophobia or the inability to lie still in a confined space
* physical disabilities that prohibit task performance (e.g., blindness or deafness)
* positive pregnancy test
* cochlear implant
* an implanted neurostimulator
* physical disabilities that prohibit task performance (e.g., blindness or deafness)
* vulnerable populations (i.e., pregnant women, individuals appearing to lack consent capacity, prisoners, individuals unable to read consent materials, individuals in a relationship with study researchers (e.g., friends, family members, significant others)
* having a history of chest pain during physical activity
* having a bone, joint, cardiac, or other medical condition that a doctor has said may be worsened by physical activity
* having asthma
* responding 'Yes' to any of the seven questions on the Physical Activity Readiness Questionnaire (PAR-Q - administered as part of the Exercise Safety Questions of the phone screen), indicating it is unsafe for the individual to engage in aerobic exercise without physician approval (i.e., potential participant would be eligible to participate if they indicated 'Yes' to one or more of the PAR-Q items provided they obtain a doctor's note indicating it is safe for them to participate in the study)
* Percutaneous Coronary Intervention or acute myocardial infarction in the last 6 weeks
* unstable arrhythmias/implanted cardiac defibrillator shocks in the last 3 months
* any other condition that the PI believes might put the participant at risk.
* Additionally, due to their effects on image quality, interested individuals with the following may be ineligible to participate per PI's judgement: nonremovable dental implants (e.g., braces or upper permanent retainers) as these will distort the MRI images we collect (note: filings, crowns, and silver or gold teeth are okay); any other condition, medication, or implant that the PI believes would degrade image quality or render data unusable

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Skin conductance responses | Collected during fear conditioning, fear extinction, and extinction recall task.
  SCR data will be collected while participants are completing the cognitive task in the MRI environment.
Threat expectancy ratings | Collected during fear conditioning, fear extinction, and extinction recall task.
  Threat expectancy ratings will be collected while participants are completing the cognitive task in the MRI environment.
Neural activity | Collected during fear conditioning, fear extinction, and extinction recall task.
  Neural activity will be collected while participants are completing the cognitive task in the MRI environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Wade Hall - University of Alabama, Tuscaloosa, Alabama, United States